CLINICAL TRIAL: NCT03818971
Title: Study of Retinal Function Using Electroretinogram in Regular Alcohol Users
Acronym: ERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RIPH 2018-02; IDRCB 2018-A02336-49 (Other: ANSM (French competent authority))
Record Dates: First submitted 2019-01-10; First posted 2019-01-28 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Use Disorder
Keywords: retina AND electroretinogram
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: mono centric study, in parallel groups, controlled, non-randomized and open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- alcohol consumption with alcohol use disorder (AUD) (Experimental): subjects with regular alcohol consumption with AUD according to the DSM 5 without any other substance use disorder (except alcohol) without psychiatric, neurologic or ophthalmologic disease in progress with a negative drug check and Breathalyzer the day of the inclusion - only one visit is planned for this study : an electroretinogram will be realized
  Interventions: Other: electroretinogram (flash, pattern and multifocal)
- alcohol consumption without alcohol use disorder (Other): subjects with regular alcohol consumption without AUD according to the DSM 5 without any other substance use disorder without psychiatric, neurologic or ophthalmologic disease in progress with a negative drug check and Breathalyzer the day of the inclusion - only one visit is planned for this study : an electroretinogram will be realized
  Interventions: Other: electroretinogram (flash, pattern and multifocal)
- no alcohol consumption (Other): subjects without alcohol consumption without any other substance use disorder without psychiatric, neurologic or ophthalmologic disease in progress with a negative drug check and Breathalyzer the day of the inclusion - only one visit is planned for this study : an electroretinogram will be realized
  Interventions: Other: electroretinogram (flash, pattern and multifocal)

INTERVENTIONS:
Other: electroretinogram (flash, pattern and multifocal) — we measured the waves a, b, oscillatory potentials, back ground noise and i for the flash ERG, the waves P50 and N95 for the pattern ERG and the P1, N1 and N2 for the multifocal ERG

SUMMARY:
Alcohol is a major public health problem and its neurotoxic effects are, among other things, responsible for altering the functioning of cerebral neurotransmission pathways.

The retina is an anatomical and developmental extension of the central nervous system. It is composed of several layers of retinal neurons that share similar anatomical and functional properties with brain neurons. Retinal neurons are notably equipped with a complex system of neurotransmission constituted by the main neurotransmitters that are involved in the central effects of alcohol: glutamate, dopamine, serotonin ... The retina is used here as a site of indirect investigation for abnormal central neurotransmission pathways following regular alcohol use. It is recognized to date as a good site for investigating central abnormalities in neuropsychiatric and addictive disorders.

The objective of this project is to study the retinal function using electroretinogram (ERG) in regular alcohol users to isolate potential markers of cerebral neurotransmission abnormalities.

ELIGIBILITY:
For alcohol consumer with alcohol use disorder :

Inclusion Criteria:

* aged between 18 and 35 years
* alcohol use disorder according to the DSM 5
* affiliation to a social security scheme

Exclusion Criteria:

* psychoactive substance consumption (other than alcohol)
* psychiatric disease in progress according to the DSM 5
* neurologic disease in progress
* mental impairment making it difficult or impossible to participate to the study
* major under guardianship or curatorship or under safeguarding of justice
* pregnant women or feeding
* people in emergency situation
* participation to another interventional study
* retinal disease in progress
* chronic glaucoma
* ophtalmic disease affecting the visual acuity
* ocular infection in progress
* urinary positive drug check the day of the inclusion
* postive Breathalyser the day of the inclusion

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
modification of amplitude | Day 0 (=day of inclusion = the only visit of the study)
  measured with flash electroretinogram and pattern electroretinogram / amplitude in microvolt
modification of implicite time parameters | Day 0 (=day of inclusion = the only visit of the study)
  measured with flash electroretinogram and pattern electroretinogram - implicite time in millisecond
modification of amplitude of the oscillatory potential | Day 0 (=day of inclusion = the only visit of the study)
  waves P1, P2, P3, P4 measured with flash electroretinogram - amplitude in microvolt
modification of implicit time of the oscillatory potential | Day 0 (=day of inclusion = the only visit of the study)
  waves P1, P2, P3, P4 measured with flash electroretinogram - implicite time in millisecond
modification of amplitude of the background noise | Day 0 (=day of inclusion = the only visit of the study)
  measured with the flash electroretinogram, flicker 3.0 sequence - amplitude in microvolt

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SCHWITZER, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, Nancy, France

IPD SHARING:
Plan to Share IPD: No